CLINICAL TRIAL: NCT04843488
Title: Effectiveness of Different Membrane Applications (Perforated Polytetrafluroethylene (PTFE) vs. Perforated PTFE+ Collagen Membrane) in Vertical Ridge Augmentation - Randomized Clinical Trial
Brief Title: Effectiveness of Different Membrane Applications in Vertical Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urban Regeneration Institute (Other)
Collaborators: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTFE1
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-06

CONDITIONS: Bone Regeneration; Dental Implants; Polytetrafluoroethylene
Keywords: Guided Bone Regeneration; Vertical Ridge Regeneration; PTFE membrane

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ridge Augmentation with a perforate PTFE mesh (Active Comparator): Vertical and horizontal ridge augmentation will be performed using d-PTFE mesh. The graft material is autograft mixed with a xenograft in a 1:1 ratio.
  Interventions: Procedure: Guided bone regeneration with a PTFE membrane
- Ridge Augmentation with a perforate PTFE mesh covered with a collagen membrane (Experimental): Vertical and horizontal ridge augmentation will be performed using d-PTFE mesh. The mesh will be covered with a native collagen membrane. The graft material is autograft mixed with a xenograft in a 1:1 ratio.
  Interventions: Procedure: Guided bone regeneration with a PTFE+collagen membrane

INTERVENTIONS:
Procedure: Guided bone regeneration with a PTFE membrane — Xenograft bovine spongious bone substitute mixed with autogenous intraorally harvested particulated bone is used and spatially contained with a PTFE membrane secured with Ti pins and screws.
  Arms: Ridge Augmentation with a perforate PTFE mesh
Procedure: Guided bone regeneration with a PTFE+collagen membrane — Xenograft bovine spongious bone substitute mixed with autogenous intraorally harvested particulated bone is used and spatially contained with a PTFE membrane secured with Ti pins and screws and covered with a Collagen membrane subsequently.
  Arms: Ridge Augmentation with a perforate PTFE mesh covered with a collagen membrane

SUMMARY:
This randomized clinical trial (RCT) study investigates if there is any difference in absolute vertical bone gain between perforated dense-polytetrafluroethylene (d-PTFE) mesh vs perforated d-PTFE mesh covered with a native collagen membrane.

The primary endpoint is absolute vertical bone gain. The secondary endpoints are regeneration rate, complications rate, and pseudoperiosteum formation.

ELIGIBILITY:
Inclusion Criteria:

1. Partially edentulous patients requiring vertical and horizontal ridge augmentation
2. patients agrees with conditions of the study and sign consent

Exclusion Criteria:

* Insufficient oral hygiene
* Smoking
* Alcohol or Drug abuse
* acute local or systemic infections
* uncontrolled diabetes or other metabolic disease
* severe hepatic or renal disfunction
* autoimmune disease
* radiotherapy in the last 5 years
* patients receiving immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Complication rate | 9 months
  intrasurgical complications such as flap perforation, mesh exposure, postoperative infection, neurosensory disturbance,
Bone gain | 9 months
  Vertical and horizontal bone gain measured

CONTACTS AND LOCATIONS:
Locations (1):
- Urban Regeneration Institute, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urban IA, Montero E, Monje A, Sanz-Sanchez I. Effectiveness of vertical ridge augmentation interventions: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:319-339. doi: 10.1111/jcpe.13061. PMID 30667522
- [Background] Urban IA, Monje A, Lozada J, Wang HL. Principles for Vertical Ridge Augmentation in the Atrophic Posterior Mandible: A Technical Review. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):639-645. doi: 10.11607/prd.3200. PMID 28817126
- [Background] Plonka AB, Urban IA, Wang HL. Decision Tree for Vertical Ridge Augmentation. Int J Periodontics Restorative Dent. 2018 Mar/Apr;38(2):269-275. doi: 10.11607/prd.3280. PMID 29447321
- [Background] Urban IA, Monje A, Lozada JL, Wang HL. Long-term Evaluation of Peri-implant Bone Level after Reconstruction of Severely Atrophic Edentulous Maxilla via Vertical and Horizontal Guided Bone Regeneration in Combination with Sinus Augmentation: A Case Series with 1 to 15 Years of Loading. Clin Implant Dent Relat Res. 2017 Feb;19(1):46-55. doi: 10.1111/cid.12431. Epub 2016 May 30. PMID 27238406
- [Background] Urban IA, Monje A, Nevins M, Nevins ML, Lozada JL, Wang HL. Surgical Management of Significant Maxillary Anterior Vertical Ridge Defects. Int J Periodontics Restorative Dent. 2016 May-Jun;36(3):329-37. doi: 10.11607/prd.2644. PMID 27100802
- [Derived] Urban IA, Serroni M, Dias DR, Barath Z, Forster A, Araujo TG, Saleh MHA, Cucchi A, Ravida A. Impact of Collagen Membrane in Vertical Ridge Augmentation Using Ti-Reinforced PTFE Mesh: A Randomised Controlled Trial. J Clin Periodontol. 2025 Apr;52(4):575-588. doi: 10.1111/jcpe.14129. Epub 2025 Feb 14. PMID 39953742